CLINICAL TRIAL: NCT00799773
Title: STAR - Study of TTP and Rituximab, A Randomized Clinical Trial
Brief Title: Evaluating the Effectiveness of Adding Rituximab to Standard Treatment for Thrombotic Thrombocytopenic Purpura (TTP)
Acronym: STAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 558; U01HL072268 (NIH); HL072268; HL072033; HL072291; HL072196; HL072248; HL072191; HL072305; HL072028; HL072072; HL072355; HL072283; HL072346; HL072331; HL072290
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Thrombotic Thrombocytopenic Purpura
Keywords: TTP; Rituximab; Plasma Exchange
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Rituximab; Plasma Exchange; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive rituximab in addition to plasma exchange and corticosteroids.
  Interventions: Drug: Rituximab; Procedure: Plasma exchange; Drug: Corticosteroids
- 2 (Active Comparator): Participants will receive plasma exchange and corticosteroids.
  Interventions: Procedure: Plasma exchange; Drug: Corticosteroids

INTERVENTIONS:
Drug: Rituximab — Dose of 375 mg/m2, given intravenously, repeated at 1-week intervals for a total of four doses
  Other Names: Rituxan
  Arms: 1
Procedure: Plasma exchange — Target volume of 1.25 plasma volume replacement; fresh frozen plasma (FFP) is the required replacement fluid; provided daily until platelet counts are normal and signs of tissue damage have improved.
Drug: Corticosteroids — 1 mg/kg of prednisone (or equivalent) each day until plasma exchange is stopped

SUMMARY:
Thrombotic thrombocytopenic purpura (TTP) is a rare disorder that causes blood clots to form in blood vessels. The main treatment for TTP is plasma exchange, in which affected patients receive transfusions of plasma, the liquid part of blood, from healthy donors. This study will examine the effectiveness of an antibody, rituximab, in combination with plasma exchange, at improving the immune response in people with TTP and decreasing the recurrence of TTP.

DETAILED DESCRIPTION:
TTP is a disorder that causes blood clots to form in the small blood vessels throughout the body. If the clots in fact block the blood vessels, blood flow is restricted to various organs, including the brain, kidneys, and heart. This can lead to neurological problems, stroke, abnormal kidney function, and heart problems. Because a large number of platelets are used in the blood clotting process, people with TTP have a reduced number of platelets circulating in their blood. They also have fewer red blood cells circulating in their blood because the red blood cells break down prematurely as blood squeezes past a blood clot.

The primary treatment for TTP is plasmapheresis, also called plasma exchange, which is a procedure that circulates a person's blood through a machine that first removes the damaged plasma and then adds healthy donor plasma into the blood. Next, patients receive a blood transfusion with the new blood. Corticosteroids, a type of medication that reduces the amount of antibodies a person's body makes, are also commonly used in conjunction with plasma exchange to treat TTP. Plasma exchange is usually effective, with platelet and red blood cell counts returning to normal after the procedure is complete. However, some people do experience a relapse of TTP and will require repeat plasma exchanges. Rituximab, an antibody currently used to treat lymphoma and rheumatoid arthritis, may improve immune system response and decrease the number of days needed to undergo the plasma exchange procedure. The purpose of this study is to evaluate the effectiveness of rituximab in combination with plasma exchange at improving an early treatment response in people with TTP and decreasing the likelihood of a relapse of TTP.

This 3-year study will enroll people who have recently been diagnosed with TTP or recently experienced a relapse and have not yet had six plasma exchanges during the current episode of TTP. Participants will be randomly assigned to receive either plasma exchanges and corticosteroids or plasma exchanges, corticosteroids, and rituximab. Blood will be collected from participants at baseline and each day they undergo the plasma exchange procedure. All participants will receive a plasma exchange every day until their platelet counts are normal and signs of tissue damage have improved. Participants will receive corticosteroid medication every day until plasma exchange is stopped, at which time the dosage will be gradually tapered until 7 weeks after the last plasma exchange. Participants receiving rituximab will receive the first dose intravenously within 7 days of the first plasma exchange; they will continue to receive rituximab once a week for 4 weeks. After the plasma exchanges are completed, all participants will have routine follow-up care with their doctors to make sure there is no TTP relapse. In the 1 year after study entry, additional blood collections will occur at varying times. Study researchers will monitor participants' health in the 3 years after study entry by following up with their doctors or through periodic phone calls. A portion of blood will be collected and stored for future TTP research purposes; this is optional.

ELIGIBILITY:
Inclusion Criteria:

* Differential or admission diagnosis of TTP-like syndrome, defined as the following:

  1. Platelet count of less than 80,000/µL for newly diagnosed patients and less than 120,000/µL for relapsed patients
  2. Microangiopathic hemolytic anemia (MHA) with red blood cell fragmentation
  3. Lactate dehydrogenase (LDH) level greater than two times the upper limit of normal for newly diagnosed patients and greater than the upper limit of normal for relapsed patients
* Receiving or will receive treatment for TTP with plasma exchange
* Has not started the sixth plasma exchange in the current TTP episode

Exclusion Criteria:

* Treated for TTP in the 2 months before study entry
* Previously enrolled in this study
* Severe active infection indicated by sepsis (requirement for pressors with or without positive blood cultures) or clinical evidence of enteric infection with E. coli 0157 or related organism
* Currently under treatment for cancer or has a current diagnosis of cancer (other than localized skin carcinoma)
* Microangiopathic hemolytic anemia due to a mechanical heart valve
* Severe high blood pressure, as defined by systolic blood pressure of greater than 180 and diastolic blood pressure of greater than 120, or papilledema
* Has ever had an organ or stem cell transplant
* Has received calcineurin inhibitors (e.g., sirolimus, tacrolimus, cyclosporin A) in the 6 months before TTP diagnosis
* Diagnosis of disseminated intravascular coagulation (DIC), defined as the following:

  1. International normalized ratio (INR) level greater than 2.0 (unrelated to anticoagulation, unresponsive to vitamin K administration) OR
  2. Fibrinogen less than 100 mg/dL
* Pregnant
* Requires ventilator assistance or intravenous pressors for treatment of TTP. If no longer required prior to study entry, patient is eligible for the study.
* Known congenital TTP or family history of TTP
* Established diagnosis of lupus, and/or actively treated for lupus in the 60 days before study entry. In addition, people with two or more of the following systemic lupus erythematosus (SLE) clinical criteria in the 60 days before study entry will be excluded:

  1. Characteristic skin rash, either malar or photosensitive
  2. Symmetric polyarthritis
  3. Serositis, either pleurisy or pericarditis
* Previously received rituximab
* Has taken the following drugs known to be associated with TTP-like syndrome in the 3 months before study entry: clopidogrel (Plavix), ticlopidine (Ticlid), or quinine
* Will receive more than 1.5 plasma volumes per day after study entry
* HIV history or positive serology
* History of hepatitis B or positive serology for HBsAg or Anti-hepatitis B core antigen (Anti-HBc)
* History of hepatitis C
* Known persistent or unexplained platelet count below 150,000/µL in the 3 months before current TTP episode
* Known hypersensitivities or allergies to murine and/or humanized antibodies
* Currently participating in trials of investigational therapies or devices (other than investigational central catheters)
* Has ever had a diagnosis of ventricular tachycardia
* Acute transmural heart attack during the current hospital admission

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan F. Assmann, PhD, Principal Investigator — New England Research Institutes, Inc.; Jan McFarland, MD, Principal Investigator — Froedtert Hospital; Eliot Williams, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Keith McCrae, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Ellis Neufeld, MD, Principal Investigator — Boston Children's Hospital; James Bussel, MD, Principal Investigator — Weill Medical Colllege, Cornell University; Thomas Ortel, MD, Principal Investigator — Duke University; Christopher Hillyer, MD, Principal Investigator — Emory University; Paul Ness, MD, Principal Investigator — Johns Hopkins University; David Kuter, MD, Principal Investigator — Massachusetts General Hospital; Sherrill Slichter, MD, Principal Investigator — University of Washington Medical Center/Fred Hutchinson Cancer Research Center (FHCRC); Cindy Leissinger, MD, Principal Investigator — Tulane University; Ronald Strauss, MD, Principal Investigator — University of Iowa; John Hess, MD, Principal Investigator — University of Maryland; Mark Brecher, MD, Principal Investigator — University of North Carolina, Chapel Hill; James George, MD, Principal Investigator — University of Oklahoma; Barbara Konkle, MD, Principal Investigator — University of Pennsylvania; Darrell Triulzi, MD, Principal Investigator — University of Pittsburgh Presbyterian and Shadyside/Children's Hospital Pittsburgh; Joseph Kiss, MD, Study Chair — University of Pittsburgh
Locations (23):
- United States (23):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital Cleveland, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Pittsburgh Presbyterian and Shadyside Hospital, Pittsburgh, Pennsylvania
  - Puget Sound Blood Center, Seattle, Washington
  - Gunderson Clinic, LTD, La Crosse, Wisconsin
  - University of Wisconsin at Madison, Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Participants will receive rituximab in addition to plasma exchange and corticosteroids.
- Standard of Care: Participants will receive plasma exchange and corticosteroids.
Period: Overall Study
Arm/Group | Rituximab | Standard of Care
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Standard of Care | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.5 (26.2) | 24 | 37 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Role of Rituximab in Increasing Early Treatment Response in Participants With TTP Who Are Also Treated With Plasma Exchange and Corticosteroids
Time Frame: Measured at Day 52
Population: The STAR informed consent form told subjects their data would be combined with other subjects' data in study reports. Because one treatment arm included only one subject, this subject's data cannot be combined with other subjects' data. Therefore, to protect subject confidentiality, results are not being released for this study.
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Use of Non-study Treatment
Time Frame: Measured at Month 36
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Whether Participants Receiving Rituximab Achieve Early or Late Treatment Response Faster and Require Fewer Plasma Exchanges Than Participants Not Receiving Rituximab
Time Frame: Measured at Days 52 and 82
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Relationship Between Clinical and Laboratory Data and Response to Treatment
Time Frame: Measured at Days 52 and 82
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Relapse Among Participants in the Two Study Groups Who Achieve Early Treatment Response
Time Frame: Measured at Month 36
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: All Cause Mortality
Time Frame: Measured at Month 36
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Treatment-related Complications
Time Frame: Measured at Day 52
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Evaluating How Levels of ADAMTS-13 Enzyme and Autoantibody at Specific Time Points or Over the Course of the Study Correlate With Other Indicators of Disease Activity, Remission Rates, Rapidity of Achieving a Remission, and Recurrence Rate
Time Frame: Measured at Month 36
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Rituximab Response in Participants With Varying Levels of ADAMTS-13 Activity and Antibodies Against ADAMTS-13
Time Frame: Measured at Month 36
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Effect of Plasma Exchange on Rituximab Levels
Time Frame: Measured at Month 6
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Effect of Rituximab Levels on the Extent of B-cell Depletion (CD-19+ Cells)
Time Frame: Measured at Month 12
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: B-cell Depletion in Relation to ADAMTS-13 Activity and to ADAMTS-13 Antibody Levels and Disease Activity in Participants Who Receive Rituximab Versus Those Who do Not
Time Frame: Measured at Month 12
Population: as for outcome 1
Arm/Group | Rituximab | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The STAR informed consent form told subjects their data would be combined with other subjects' data in study reports. Because one treatment arm included only one subject, to protect subject confidentiality adverse events, though collected, are not being reported for this study.
Arm/Group | Rituximab | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
One treatment arm had only one subject, so to protect patient confidentiality, results are not being entered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No